CLINICAL TRIAL: NCT07359105
Title: A Registry-based Randomized Controlled Trial of Moderate-intensity Statin Therapy vs. Individualized Low-density Lipoprotein Cholesterol Target-based Therapy for Primary Prevention of Cardiovascular Events in Patients 70 Years of Age or Older With Type 2 Diabetes (iTARGET-Elderly Study)
Brief Title: Moderate-intensity Statin vs. Individualized LDL-C Target-based Therapy in Older Adults With Type 2 Diabetes (iTARGET-Elderly Study)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sin Gon Kim (Other)
Collaborators: Severance Hospital (Other); Hanmi Pharmaceutical Company Limited (Industry); Yuhan Corporation (Industry)
Responsible Party: Sponsor-Investigator, Sin Gon Kim, Professior, Department of Endocrinology and metabolism, Korea University Anam Hospital, South Korea, Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025AN0165
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Dyslipidemia; T2D; Diabetes; Statins; iTARGET-Elderly; RRCT
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus | interventions — Ezetimibe

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned in a 1:1 ratio at Visit 1, using the Interactive Web Response System (IWRS), to either the moderate-intensity statin monotherapy arm or the individualized LDL-C target-based therapy arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-intensity statin monotherapy arm (Active Comparator): Statin monotherapy with approved medications.
  Interventions: Drug: Moderate-intensity statin monotherapy
- Individualized LDL-C target-based therapy arm (Experimental): The investigator will establish individualized LDL-C targets (<55 mg/dL or <70 mg/dL or <100 mg/dL) by considering each patient's cardiovascular risk, life expectancy, risk of adverse drug reactions, comorbidities, and personal preferences. The decision-making process will be shared with the patient to ensure that individual needs are addressed.
  Interventions: Drug: Ezetimibe or ezetimibe-statin combination therapy

INTERVENTIONS:
Drug: Moderate-intensity statin monotherapy — Atorvastatin 10 mg, 20 mg, or 40 mg, or rosuvastatin 5 mg, 10 mg, or 20 mg will be administered for up to 3 years. If the LDL-C is ≥100 mg/dL, the investigator may adjust the statin intensity based on the patient's health status.
  Arms: Moderate-intensity statin monotherapy arm
Drug: Ezetimibe or ezetimibe-statin combination therapy — Treatment will consist of non-pharmacological interventions or marketed medications, including low-dose statins (atorvastatin 5 mg or 10 mg, rosuvastatin 2.5 mg or 5 mg) in combination with ezetimibe 10 mg, or fixed-dose combinations (rosuvamibe 10/2.5 mg, atorvabmibe 10/5 mg, or Rosuzet 10/2.5 mg), for up to 3 years. If the pre-specified LDL-C target is not achieved or drug intolerance occurs, adjustments in dosage or medication will be made.
  Arms: Individualized LDL-C target-based therapy arm

SUMMARY:
Statins are the cornerstone of cardiovascular disease (CVD) prevention through the lowering of low-density lipoprotein cholesterol (LDL-C). While the benefits of intensive LDL-C lowering are well-established for secondary prevention, evidence remains insufficient for primary prevention in the elderly-specifically for individuals aged 70 years or older with type 2 diabetes who have no prior history of atherosclerotic cardiovascular events.

Current guidelines generally recommend moderate-intensity statins for this population based on extrapolated data. However, there is a significant evidence gap regarding whether these older adults, who have not yet experienced a cardiovascular event, derive the same risk-benefit ratio from pharmacological intervention as younger or secondary prevention groups. Furthermore, while ezetimibe (alone or in combination) is an effective alternative for patients with established disease, its efficacy as a primary prevention strategy in older diabetic patients has not been rigorously confirmed through randomized controlled trials (RCTs).

Therefore, this study specifically focuses on the primary prevention setting, aiming to determine whether individualized LDL-C target-based therapy is non-inferior to standard moderate-intensity statin therapy in preventing first-time cardiovascular events among older patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent to participate in the study by the patient or his/her legally authorized representative after receiving and understanding a detailed explanation of the study
* Adults aged 70 years or older
* Diagnosed with type 2 diabetes or currently receiving antidiabetic medication, without a history or presence of cardiovascular disease
* Either: (1) LDL-C≥100 mg/dL if not receiving lipid-lowering therapy, or (2) currently receiving lipid-lowering therapy (in this case, LDL-C level not restricted)

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Documented history of atherosclerotic cardiovascular disease at screening, confirmed clinically or by imaging: (1) myocardial infarction; (2) coronary revascularization; (3) currently receiving treatment for acute coronary syndrome; (4) history of ischemic stroke; (5) aortic aneurysm; (6) peripheral arterial disease
* Currently undergoing cancer treatment
* Severe disease requiring recurrent hospitalization
* Frailty (defined as a score ≥3 on the Korean FRAIL questionnaire), or any condition significantly limiting self-care
* AST or ALT >3 × ULN, at screening (however, patients will be eligible if repeat testing at the time of randomization shows levels <3 × ULN), or liver cirrhosis
* Contraindications to study drugs
* Pregnant or breastfeeding women

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 2186 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from the date of randomization to the first occurrence of a major adverse cardiovascular event (MACE) | 0, 3, 12, 24, 36 months
  Major adverse cardiovascular event (MACE) includes death from cardiovascular causes, non-fatal myocardial infarction, non-fatal stroke, hospitalization due to heart failure, coronary revascularization, or all-cause death.

SECONDARY OUTCOMES:
Time from the date of randomization to the first hospitalization due to the following events or to the first occurrence of such events, whichever occurs earlier : (1) ischemic heart disease, (2) cerebrovascular disease, (3) heart failure, (4) peripheral | 0, 3, 12, 24, 36 months
Time from the date of randomization to the first occurrence of all-cause hospitalization or all-cause death, whichever occurs first | 0, 3, 12, 24, 36 months
Serum lipid levels from baseline at each assessment time point | 0, 3, 12, 24, 36 months
Serum lipid changes from baseline at each assessment time point | 0, 3, 12, 24, 36 months
Patterns of study drug use | From baseline up to 36 months
Incidence rates and characteristics of adverse events, adverse drug reactions, and serious adverse events | From baseline up to 36 months
Incidence rates and characteristics of adverse events of special interest (AESI) | From baseline up to 36 months
  Adverse events of special interest (AESI): (1) Elevation of aminotransferase levels, (2) Rhabdomyolysis/myopathy, (3) Gastrointestinal problems

CONTACTS AND LOCATIONS:
Overall Officials: Sin Gon Kim, MD, Principal Investigator — Korea University Anam Hospital; Bong-Soo Cha, MD, Principal Investigator — Severance Hospital
Locations (2):
- South Korea (2):
  - Korea University ANAM Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No